CLINICAL TRIAL: NCT03937414
Title: The Validation Study of the Intraoperative OSNA Molecular Assay
Brief Title: Intraoperative Molecular Diagnosis of Sentinel Lymph Node In Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Direct of Breast Cancer Center, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSNA
Record Dates: First submitted 2019-04-27; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Sentinel Lymph Node Biopsy
Keywords: Breast neoplasm; Molecular Diagnostic Techniques
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- SLNs were tested by the OSNA assay Intraoperatively (Experimental): SLNs were tested by the OSNA assay Intraoperatively
  Interventions: Device: The OSNA assay

INTERVENTIONS:
Device: The OSNA assay — SLN was defatted after SLNB. If the node weighed less than 100mg, the node was only assessed by histology postoperatively. If the node weighed more than 100mg, the node was sliced to equal blocks according to the length of short axis: If the length was less than 4mm, the node was sliced into two blocks along the long axis (a, b). Intraoperatively, the block a and b were tested by TIC, and the block a was prepared for OSNA. Postoperatively, the block b was assessed by histology. If the length was more than 4mm, the node was sliced into four blocks (a, b, c, d). Intraoperatively, all blocks (a, b, c, d) were tested by TIC, and the block a and c were prepared for OSNA.

SUMMARY:
One-step Nucleic Acid Ampliﬁcation assay (the OSNA assay) (Sysmex, Kobe, Japan) was an objective molecular technique that combines node tissue homogenization and subsequent reverse-transcription loop-mediated isothermal ampliﬁcation of CK-19 mRNA in a single quick step. In the study, the performance of the OSNA assay was compared with the present standard histological evaluation, and a comparative analysis of OSNA assay with Touch Imprint Cytology (TIC) was also been made.

DETAILED DESCRIPTION:
Patients:

More than 1000 consecutive breast cancer patients scheduled for Sentinel Lymph Node Biopsy (SLNB) were enrolled in the study. The study was approved by the ethics committee of each center and each patient provided informed consent. The patients who had undergone previous ipsilateral axillary surgery were excluded from this study.

Sampling method:

Sentinel Lymph Node (SLN) was defatted after SLNB. If the node weighed less than 100mg, the node was only assessed by histology postoperatively. If the node weighed more than 100mg, the node was sliced to equal blocks according to the length of short axis: If the length was less than 4mm, the node was sliced into two blocks along the long axis (a, b). Intraoperatively, the block a and b were tested by TIC, and the block a was prepared for OSNA. Postoperatively, the block b was assessed by histology. If the length was more than 4mm, the node was sliced into four blocks (a, b, c, d). Intraoperatively, all blocks (a, b, c, d) were tested by TIC, and the block a and c were prepared for OSNA. Postoperatively, the block b and d were subjected to histology. ALND was only performed if the TIC results were positive.

OSNA assay:

All the assay operators attended a three-day-training course before the study. OSNA assay was performed according to the manufacturer's instructions. Three different calibrators with defined CK-19 mRNA copy concentrations were used to construct a standard curve on Sysmex RD-100i instrument. Then, node tissues were homogenized in 4ml homogenizing buffer Sysmex LYNORHAG. Afterwards, the homogenate was briefly centrifuged and directly used as a template for RT-LAMP. Amplification of CK-19 mRNA was automatically performed in SysmexTM RD-100i instrument with a ready-to-use reagent Sysmex LYNOAMP kit which consists of a primer-nucleotide-mix, enzymes and CK-19 mRNA calibrators as well as positive and negative controls. All the results were presented on the RD-100i instrument in qualitative categories [++, +, -] and further specified by CK-19 mRNA copy number/μl: ~250 copies [-], 250~5000 copies [+], and 5000~ [++]. The result [+] was comparable to the presence of a micro-metastasis, and [++] to a macro-metastasis.

Histological evaluation:

All node blocks used for histological evaluation were fixed in 10% buffered formalin and paraffin embedded. Four 4~6μm thick slides 200μm apart were taken from each block. Metastases larger than 0.2mm were considered positive in this study. Metastases were classified according to the 7th criterion of American Joint Cancer Committee. Macro-metastases (≥2mm) and micro-metastases (0.2~2mm, pT1mic) were considered node positive. Isolated tumor cells [≤0.2mm, ITCs, pT0(i+)] were considered node negative. All the slides were reviewed by a senior pathologist from another center. When there was a disagreement, a third senior pathologist was attended to make the final diagnosis. All the pathologists were blinded to the OSNA results.

Statistical methods:

The primary goal was the accuracy, sensitivity, specificity of the OSNA assay. McNemar test was performed to compare the rate between groups.

ELIGIBILITY:
Inclusion Criteria:

The breast cancer patients scheduled for SLNB.

Exclusion Criteria:

The patients who had undergone previous ipsilateral axillary surgery.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2010-02-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The accuracy, sensitivity, specificity of the OSNA assay | 10 years
  The accuracy, sensitivity, specificity of the OSNA assay

CONTACTS AND LOCATIONS:
Overall Officials: Yong-sheng Wang, Principal Investigator — Shandong Cancer Hospital & Institute
Locations (1):
- Breast Cancer Center, Shandong Cancer Hospital Affiliated to Shandong University, Jinan, China

REFERENCES:
- [Result] Wang YS, Ou-yang T, Wu J, Liu YH, Cao XC, Sun X, Fu L, Liao N, Yang WT, Zhong WX, Lu AP. Comparative study of one-step nucleic acid amplification assay, frozen section, and touch imprint cytology for intraoperative assessment of breast sentinel lymph node in Chinese patients. Cancer Sci. 2012 Nov;103(11):1989-93. doi: 10.1111/cas.12001. Epub 2012 Oct 18. PMID 22924886